CLINICAL TRIAL: NCT01132456
Title: RESOLUTE Asia: Evaluation of the Endeavor Resolute Zotarolimus-Eluting Coronary Stent System in a Patient Population With Long Lesion(s) and/or Dual Vessels in Asia
Brief Title: RESOLUTE Asia: Evaluation of the Endeavor Resolute Zotarolimus-Eluting Stent System in a Patient Population With Long Lesion(s) and/or Dual Vessels in Asia
Acronym: R-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP123
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Ischemic Heart Disease; Coronary Stenosis; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease
Keywords: TARGET VESSEL REVASCULARIZATION (TVR); MYOCARDIAL INFARCTION (MI); TARGET VESSEL FAILURE (TVF); TARGET LESION REVASCULARIZATION (TLR); TARGET LESION FAILURE (TLF); STENT THROMBOSIS; RESTENOTIC LESION; PERCUTANEOUS CORONARY INTERVENTION (PCI); LONG LESION; DUAL VESSEL
MeSH Terms: conditions — Myocardial Ischemia; Coronary Stenosis; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Different patient subset (Experimental): Patients with dual vessel treatment where each vessel has a lesion with length ≤ 27 mm and reference vessel diameters between 2.25 mm and 4.0 mm.
  Interventions: Device: Drug eluting stent treatment
- 38 mm Cohort (Experimental): Patients with at least one lesion amenable to treatment with a 38 mm length Endeavor Resolute stent. Patients may have one or two lesions, if the two lesions are located in separate target vessels.
  Interventions: Device: Drug eluting stent treatment

INTERVENTIONS:
Device: Drug eluting stent treatment — Endeavor RESOLUTE Zotarolimus-Eluting Coronary Stent Implantation

SUMMARY:
The purpose of this study is to document the safety and overall clinical performance of the Endeavor Resolute Zotarolimus-Eluting Coronary Stent System in a patient population with long lesion(s) and/or dual vessels requiring stent implantation.

DETAILED DESCRIPTION:
A total of 249 to 411 patients will be enrolled from Asia at approximately 25 centers where Endeavor Resolute stent is commercially available. There are two study cohorts:

1. 38 mm cohort: a minimum of 46 patients and maximum of 111 patients with at least one lesion amenable to treatment with a 38 mm length Endeavor Resolute stent. Patients may have one or two lesions, if the two lesions are located in separate target vessels.
2. Dual vessel cohort: a minimum of 203 patients and maximum of 300 patients with dual vessel treatment where each vessel has a lesion with length ≤ 27 mm and reference vessel diameters between 2.25 mm and 4.0 mm.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable candidate for percutaneous coronary intervention (PCI),stenting, and emergency coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia and/or positive functional study
* Informed consent
* Patient agrees to comply with specified follow-up evaluations at same investigational site
* Single target lesion or two target lesions located in separate coronary arteries
* De novo lesion(s) in native coronary artery(ies)
* Target lesion(s) ≤ 35 mm in length (or both lesion lengths ≤ 27 mm for two lesions in separate target vessels to be considered for the dual vessel cohort)
* Target vessel(s) have reference vessel diameter 2.25 mm to 4.0 mm, (or 3.0 to 4.0 mm for it to be treated with a 38 mm length stent)

Exclusion Criteria:

* Within 7 days of implant platelet count <100,000 cells/mm³ or >700,000 cells/mm³; WBC count <3,000 cells/mm³; serum creatinine level >2.5 mg/dl
* Acute MI within 72 hrs of the index procedure (QWMI or any elevation of CK-MB > lab upper limit of normal)
* Previous PCI of target vessel(s) within 9 months prior to the procedure
* Planned PCI of any vessel within 30 days post-index procedure and/or planned PCI of target vessel(s) within 12 months post-index procedure
* History of stroke or TIA within prior 6 months
* Participating in investigational drug/device study that has not completed primary endpoint or interferes with study endpoints
* Inability to comply with required trial antiplatelet regimen
* Previous stent in target vessel unless it has been at least 9 months since stent placed and target lesion(s) is/are at least 15 mm from previous stent
* Target vessel(s) has/have other lesions w/ > 40% diameter stenosis
* Unprotected left main coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) for 38mm cohort and Target Vessel Failure (TVF) for dual vessel cohort | 12 months
  TLF is defined as composite of cardiac death, target vessel myocardial infarction (Q wave and non-Q wave) or clinically-driven target lesion revascularization (TLR) by percutaneous or surgical methods. TVF is defined as composite of cardiac death, target vessel myocardial infarction (Q wave and non-Q wave) or clinically-driven target vessel revascularization (TVR).

SECONDARY OUTCOMES:
Death | 30d, 6m, 9m, 12m, 18m, 2yr, 3yr
  Death rate in the study.
MI | 30d, 6m, 9m, 12m, 18m, 2yr, 3yr
  Myocardial infarction (MI) rate in the study.
Cardiac death and MI | 30d, 6m, 9m, 12m, 18m, 2yr, 3yr
  Cardiac death and myocardial infarction (MI) rate in the study
MACE | 30d, 6m, 9m, 12m, 18m, 2yr, 3yr
  MACE composite endpoint and each individual component (death, myocardial infarction (MI) (Q wave and non-Q wave), emergent coronary bypass surgery (CABG), or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods)
TLF | For 38mm cohort it is 30d, 6m, 9m, 18m, 2yr and 3yr. For dual vessel cohort it is 30d, 6m, 9m, 12m, 18m, 2yr and 3yr
  TLF composite endpoint and each individual component (cardiac death, target vessel MI or clinically-driven TLR)

CONTACTS AND LOCATIONS:
Overall Officials: Robaayah Zambahari, MBBS, MRCP, FRCP, FACC, Principal Investigator — National Heart Institute (IJN), Malaysia; Michael Kang-Yin Lee, MBBS, Principal Investigator — Queen Elizabeth Hospital, HK; Shirish Hiremath, MD, Principal Investigator — Ruby Hall Clinic, India
Locations (1):
- The Heart Care Clinic, Ahmedabad, Gujarat, India

REFERENCES:
- [Result] Lee M, Hiremath S, Zambahari R, Leon M, Mauri L, Yeung A; RESOLUTE US and RESOLUTE Asia Investigators. One-year outcomes of percutaneous coronary intervention with the 38-mm Resolute zotarolimus-eluting stent. Am J Cardiol. 2013 Nov 1;112(9):1335-41. doi: 10.1016/j.amjcard.2013.06.012. Epub 2013 Aug 14. PMID 23953695